CLINICAL TRIAL: NCT03193567
Title: Phase I Study of High Efficient Killing Cell Therapy for Advanced Non Small Cell Lung Cancer
Brief Title: Study of High Efficient Killing Cell Therapy for Advanced NSCLC
Acronym: HEART
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Shanghai Houchao Biotechnology Co., Ltd (Unknown)
Responsible Party: Principal Investigator, Hecheng Li M.D., Ph.D, Professor, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTS-005
Record Dates: First submitted 2017-06-16; First posted 2017-06-21 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HEKT cell (Experimental): Enrolled patients will receive HEKT cell injection, 10-days interval, totally 3 times.
  Interventions: Biological: HEKT cell

INTERVENTIONS:
Biological: HEKT cell — 3 cycles of HEKT cell treatment
  Other Names: High Efficient Killing Cell Therapy

SUMMARY:
The purpose of this study to preliminarily evaluate the safety and efficacy of High Efficient Killing Cell Therapy for refractory and advanced non-small cell lung cancer

DETAILED DESCRIPTION:
Patients with pathological confirmed non-small cell lung cancer with no standard treatment are enrolled. The patients fails in previous at least 2 lines of chemotherapy and 1 line of targeted therapy where applicable. This is a prospective exploratory trial.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients' age from 18 years to 70 years.
* Patients who have a life expectancy of at least 3 months.
* pathologically confirmed non-small cell lung cancer.
* failed in previous standard chemotherapy and targeted therapy.
* Karnofsky performance status 0-1.
* adequate organ functions.

Exclusion Criteria:

* Pregnant and lactating women.
* Patients with T cell lymphoma, syphilis, AIDS or combination
* Patients with highly allergic or have a history of severe allergies
* Patients with severe hepatic or renal dysfunction
* Patients with severe autoimmune disease or who is being treated with immunosuppressive agents
* Patients with severe infection not controlled or High fever
* Patients with organ transplantation or waiting for organ transplantation.
* Patients with brain metastasis
* Patients with severe coagulopathy (e.g. hemophilia)
* Patients without adequate ability to understand, sign informed consents and take part in the clinical research voluntarily.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2017-09-14 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
safety：safety index of blood, heart, lung, kidney and brain function damaged mainly during the treatment | 2 years
  Occurrence of study related adverse events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
efficacy: complete response; partial response; stable disease; progression disease; progression free survival. | 2 years
  The efficacy of the treatment is assessed according to (RECIST1.1)

OTHER OUTCOMES:
Progression free survival | 2 years
  Progression free survival is defined as the time from the day in which the patient is enrolled to the date on which tumor progresses or the date on which the patient dies for any cause.
Overall survival | 2 years
  Overall survival is defined as the time from the day in which the patient is enrolled to the date on which the patient dies for any cause.
Imaging evaluation before and after treatment | 0 day and 60 day
  the SUV index of PET-CT before cell injection and after the whole course of the treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, China